CLINICAL TRIAL: NCT04058444
Title: Implementation of ERAS Protocol for Cesarean Delivery in Clinical Center Vojvodina
Brief Title: The First ERAS Protocol for Cesarean Delivery in Serbia at the University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pujic Borislava (Other)
Responsible Party: Sponsor-Investigator, Pujic Borislava, Director of Obstetrical Anesthesia, University of Novi Sad
Organization: University of Novi Sad (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0712960805046
Record Dates: First submitted 2019-04-13; First posted 2019-08-15 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Cesarean Delivery
Keywords: cesarean delivery; ERAS protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS Group (Experimental): Perioperative management follows the ERAS (Enhanced Recovery After Surgery) protocol
  Interventions: Combination Product: ERAS protocol
- Control Group (Experimental): Perioperative management follows the conventional program
  Interventions: Combination Product: ERAS protocol

INTERVENTIONS:
Combination Product: ERAS protocol — No routine bowel preparation Antibiotics prophylaxis PONV (Postoperative Nausea and Vomiting) prophylaxis Spinal anesthesia Post- Cesarean analgesia (Acetaminophen 1g IV q6h, Tramadol 50mg IV q6h, Quadratus lumborum Block Oral pain relief medication Pain scores every day (VAS) Hospital length of stay Patient satisfaction

SUMMARY:
This study is designed to help us with ERAS (Enhanced Recovery After Surgery) Protocol for Cesarean Delivery implementation with goal to improve patient satisfaction and decrease length of stay at hospital. This will improve patient treatment and decrease total hospital costs.

DETAILED DESCRIPTION:
ERAS assumes cooperation between obstetricians, anesthesiologists and parturient. This is the new concept because patient have an active role in the whole process. Pregnant patient receives the first information about ERAS from obstetrician and anesthesiologist before the scheduled cesarean delivery. Patient condition optimization is necessary. Antibiotic prophylaxis, no bowel preparation and arriving to the hospital on the day of surgery are basic principles. All patients are done under spinal anesthesia. DVT (Deep Venous Thrombosis) prophylaxis starts postoperatively. Early mobilization, early oral intake and urinary catheter removal on the day of surgery with multimodal analgesia is mandatory.

ELIGIBILITY:
Inclusion Criteria:

* All healthy patients from 18-45 years for scheduled Cesarean Delivery

Exclusion Criteria:

* Age younger then 18 years old and older then 45 years
* Urgent and emergent Cesarean Delivery
* Preeclampsia
* Contraindications for spinal anesthesia
* Abnormal placentation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2019-09-19 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Post-Cesarean pain scoring | Measured from postoperative day (PO) Day 0 to PO day 3 (72 hours)
  Visual Analog Scale (VAS) for pain assessment (scale from 0-10). Score 0 to 5 is satisfactory pain control. Score 6 to 10 is not a good pain control and is necessary to add medication.

SECONDARY OUTCOMES:
Hospital length of stay | PO Day 0 until time of discharge PO Day 3-4 (72-96 hours)
  Length of stay might influence on cost savings. Investigator expects discharge hospital will be on the PO day 3.
Post-partal depression development | Measured from the Cesarean Delivery to 6 weeks postoperatively
  Inadequate postoperative treatment could cause chronic pain which could be the reason for post- partal depression development. Six weeks after delivery investigator will call mothers for interview and fill the Edinburgh Postnatal Depression Scale. Score 10 and more is suspect for depression risk.

CONTACTS AND LOCATIONS:
Overall Officials: Borislava Pujic, PhD, Principal Investigator — Obstetric and Gynecology Hospital, Novi Sad, Serbia
Locations (1):
- Obstetric and Gynecology Hospital, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gamez BH, Habib AS. Predicting Severity of Acute Pain After Cesarean Delivery: A Narrative Review. Anesth Analg. 2018 May;126(5):1606-1614. doi: 10.1213/ANE.0000000000002658. PMID 29210789
- [Result] Valentine AR, Carvalho B, Lazo TA, Riley ET. Scheduled acetaminophen with as-needed opioids compared to as-needed acetaminophen plus opioids for post-cesarean pain management. Int J Obstet Anesth. 2015 Aug;24(3):210-6. doi: 10.1016/j.ijoa.2015.03.006. Epub 2015 Mar 23. PMID 25936786
- [Result] Krohg A, Ullensvang K, Rosseland LA, Langesaeter E, Sauter AR. The Analgesic Effect of Ultrasound-Guided Quadratus Lumborum Block After Cesarean Delivery: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):559-565. doi: 10.1213/ANE.0000000000002648. PMID 29135590